CLINICAL TRIAL: NCT04695548
Title: Comparison of Isometric, Concentric, Eccentric Exercise and Passive Stretching in the Reduction of Post-needling Soreness in Patients With Cranial and/or Cervical Pain Related to Myofascial Pain
Brief Title: Physiotherapy in the Reduction of Post-needling Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/43
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Dry Needling; Soreness, Muscle; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myalgia; Myofascial Pain Syndromes | interventions — Isometric Contraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Concentric contraction exercise (Experimental): After applying the dry needling technique to the upper trapezius muscle, the participant will be placed in a standing position, with the shoulders positioned in the scapular plane. A medium stiffness Theraband elastic band will be placed between the participant's ipsilateral foot on the side on which the dry needling technique was applied and the acromio-clavicular joint on the same side.The exercise will consist of raising the shoulder against the resistance of the elastic band, slowly and for 5 seconds
  Interventions: Other: Concentric contraction exercise
- Isometric contraction exercise (Experimental): After applying the dry needling technique to the upper trapezius muscle, the participant will be placed in a standing position, with the shoulders positioned in the scapular plane. A medium stiffness Theraband elastic band will be placed between the participant's ipsilateral foot on the side on which the dry needling technique was applied and the acromio-clavicular joint on the same side.The exercise will consist of raising the shoulder and maintaining the tension of the elastic band for 5 seconds
  Interventions: Other: Isometric contraction exercise
- Eccentric contraction exercise (Experimental): After applying the dry needling technique to the upper trapezius muscle, the participant will be placed in a standing position, with the shoulders positioned in the scapular plane. A medium stiffness Theraband elastic band will be placed between the participant's ipsilateral foot on the side on which the dry needling technique was applied and the acromio-clavicular joint on the same side.The exercise will consist of raising the shoulder against the resistance of the elastic band, slowly and for 5 seconds
  Interventions: Other: Eccentric contraction exercise
- Analytic passive stretching. (Experimental): After applying the dry needling technique to the upper trapezius muscle, the patient remains supine position. The analytical passive stretch of the upper trapezius will be performed only once, bringing the muscle to the limit of elastic tension perceived by the subject. The passive stretching technique will be held for 30 seconds.
  Interventions: Other: Analytic passive stretching

INTERVENTIONS:
Other: Concentric contraction exercise — The participant will be placed in a standing position, with the shoulders positioned in the scapular plane. A medium stiffness Theraband elastic band will be placed between the participant's ipsilateral foot on the side on which the dry needling technique was applied and the acromio-clavicular joint on the same side.The exercise will consist of raising the shoulder against the resistance of the elastic band, slowly and for 5 seconds
  Other Names: Muscle concentric contraction
  Arms: Concentric contraction exercise
Other: Isometric contraction exercise — The participant will be placed in a standing position, with the shoulders positioned in the scapular plane. A medium stiffness Theraband elastic band will be placed between the participant's ipsilateral foot on the side on which the dry needling technique was applied and the acromio-clavicular joint on the same side.The exercise will consist of raising the shoulder and maintaining the tension of the elastic band for 5 seconds
  Other Names: Muscle isometric contraction
  Arms: Isometric contraction exercise
Other: Eccentric contraction exercise — The participant will be placed in a standing position, with the shoulders positioned in the scapular plane. A medium stiffness Theraband elastic band will be placed between the participant's ipsilateral foot on the side on which the dry needling technique was applied and the acromio-clavicular joint on the same side.The exercise will consist of asking the participant to lower their shoulder, against the resistance of the elastic band, in a slow and controlled manner for 5 seconds.
  Other Names: Muscle eccentric contraction
  Arms: Eccentric contraction exercise
Other: Analytic passive stretching — The patient remains supine position. The analytical passive stretch of the upper trapezius will be performed only once, bringing the muscle to the limit of elastic tension perceived by the subject. The passive stretching technique will be held for 30 seconds.
  Other Names: Muscle passive stretching
  Arms: Analytic passive stretching.

SUMMARY:
Dry needling is a minimally invasive technique which generates good results and neuromuscular benefits. Its application involves a highly prevalent effect called post-needling soreness. It is defined as a residual pain, located in the incision area, with a self-limiting period of 24-72 hours, as a result of a physiological process generated by the technique.

So far, different clinical trials have been carried out to measure the effectiveness of several techniques for reducing post-needling soreness, reaching positive results. However, no studies have been found with the aim of distinguish which method is more effective for this goal; therefore, it is clear the need to continue investigating on the subject and comparing these techniques among them.

DETAILED DESCRIPTION:
Main objective. To figure out if one of the four techniques (isometric, concentric, eccentric contraction exercise and analytic passive stretching) is more effective for reducing post- needling soreness immediately, at 12, 24, 48 and 72 hours.

Objectives. To verify if there is a correlation between independent variables and post-needling soreness.

Study type. Non-blinded randomized clinical trial. Intervention. Dry needling on an active myofascial trigger point in superior trapezius, followed by one of the following treatments according to the specific group: 1) concentric contraction exercise, 2) isometric contraction exercise, 3) eccentric contraction exercise or 4) analytic passive stretching.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Cervical pain.
* Presence of an active PGM in the upper trapezius muscle.

Exclusion Criteria:

* Traumatic history in the cervical region;
* Inability to understand or perform the required exercises;
* Pregnancy in the first trimester;
* Altered state of coagulation;
* Immunosuppression status;
* State of alteration of sensitivity (e.g. central sensitization processes, fibromyalgia, etc.);
* Unavoidable fear of needles;
* Lack of knowledge about the use of the WhatsApp or Telegram messaging platform

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Post-needling soreness intensity | Change From Baseline in Pain Scores on the Visual Analog Scale at 72 hours.
  The investigators use a Visual Analog Scale (VAS) to determine the intensity of the patient's post-needing pain after and for 72 hours after DN.The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.

SECONDARY OUTCOMES:
Pain Catastrophizing | Change from Baseline Pain Catastrophizing at 72 hours.
  This scale is a Likert-type questionnaire with 5 levels (0-4) that includes 13 items that measure 3 dimensions of catastrophism: magnification, rumination and despair. The Spanish version of this scale has shown to have an appropriate internal consistency, test-retest reliability and sensitivity to changes.
Fear of Pain. | Change from Baseline Fear of Pain at 72 hours.
  Fear of Pain Questionnaire. This scale is a Likert-type questionnaire with 5 levels (1-5) with 3 lists of 10 sub-items that contemplate 3 different aspects of fear of pain: fear of mild pain, fear of severe pain, fear of pain related to the area doctor. The Spanish version of this scale has shown to have an acceptable validity and reliability.
Pain Anxiety Symptoms | Change from Baseline Pain Anxiety at 72 hours.
  The Pain Anxiety Symptoms Scale. This Likert-type questionnaire with 6 levels (0-5) includes 20 items that measure 4 dimensions of pain anxiety: cognitive anxiety, escape / avoidance, fear and physiological anxiety. The Spanish version of this scale has been shown to have appropriate validity and reliability

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Principal Investigator — Alcala University
Locations (1):
- Clinical University Physiotherapy and pain, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No